CLINICAL TRIAL: NCT02460445
Title: Effect of Decreasing Iron Tissue Depots on the Cardiovascular Risk of Women With Polycystic Ovary Syndrome
Brief Title: Phlebotomy and Polycystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manuel Luque Ramírez (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor-Investigator, Manuel Luque Ramírez, Member of the Diabetes, Obesity and Human Reproduction Research Group, Centro de Investigación Biomédica en Red Diabetes y Enfermedades Metabólicas Asociadas CIBERDEM., Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal
Organization: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI14/00649
Record Dates: First submitted 2015-05-27; First posted 2015-06-02 (Estimated); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Hyperandrogenism; Metabolic Cardiovascular Syndrome
Keywords: Functional hyperandrogenism; Polycystic ovary syndrome; Idiopathic hyperandrogenism; Iron tissue depots; Phlebotomy; Insulin resistance; Carbohydrate metabolism; Blood pressure; Autonomic dysfunction; Oxidative stress; Blood clotting tests; Efficacy; Side effects; Randomized clinical trial
MeSH Terms: conditions — Hyperandrogenism; Metabolic Syndrome; Polycystic Ovary Syndrome; Insulin Resistance; Primary Dysautonomias | interventions — Phlebotomy; Blood Donation; Bloodletting; Ethinyl Estradiol; Cyproterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Premenopausal women with functional hyperandrogenism under combined oral contraceptive pill qd as usual clinical practice who will undergo a scheduled standard phlebotomy every 3 months from month 3 to 12 of follow-up.
  Interventions: Procedure: Phlebotomy; Drug: ethinylestradiol; Drug: Cyproterone Acetate
- Control (Active Comparator): Premenopausal women with functional hyperandrogenism under standard combined oral contraceptive pill qd as usual clinical practice.
  Interventions: Drug: ethinylestradiol; Drug: Cyproterone Acetate

INTERVENTIONS:
Procedure: Phlebotomy — Scheduled standard phlebotomy every three months from month 3 to 12 of follow-up.
  Other Names: Blood donation; Bloodletting
  Arms: Intervention
Drug: ethinylestradiol — 35 mcg ethinylestradiol qd for 21 days per month as usual clinical practice.
Drug: Cyproterone Acetate — 2 mg cyproterone acetate qd for 21 days per month as usual clinical practice.

SUMMARY:
AIMS To study the effects of the decrease in iron tissue depots after scheduled bloodletting on insulin sensitivity, carbohydrate metabolism, classic and non-classic cardiovascular risk factors in patients with functional hyperandrogenism (polycystic ovary syndrome & idiopathic hyperandrogenism) on standard treatment with combined oral contraceptives (COC) according to usual clinical practice.

METHODOLOGY

Open label, controlled, parallel, prospective study of 12 months of duration, with 2 randomized arms of follow-up:

i) Intervention Group: Patients with functional hyperandrogenism on standard COC treatment randomly allocated to perform scheduled phlebotomies from the third month of treatment to the end of the study (3 times with a 3-month interval between them).

ii) Control Group: Patients with functional hyperandrogenism on standard COC treatment randomly allocated to follow-up without bloodletting.

The whole group of patients will undergo a comprehensive anthropometric and hormonal assessment, evaluation of classic cardiovascular risk factors (insulin sensitivity and carbohydrate metabolism after a standard oral glucose test- 75 g), lipid profile, ambulatory and office blood pressure monitoring, proinflammatory profile, oxidative stress status, autonomic function assessment, and iron-related metabolism parameters at baseline, after 3-month COC treatment and after reduction of iron tissue depots plus OC in the Intervention Group of patients, and throughout follow-up under treatment with COC in the Control Group of patients. If a significant relationship between circulating hepcidin levels and elevated ferritin concentrations is observed, a study of the potential influence of mutations/polymorphic variants of hepcidin gene on ferritin values will be performed as well.

ELIGIBILITY:
Inclusion Criteria:

1. Premenopausal women with functional hyperandrogenism defined as:

   * Polycystic ovary syndrome (PCOS): Clinical and biochemical hyperandrogenism plus ovulatory dysfunction or polycystic ovarian morphology.
   * Idiopathic hyperandrogenism: Clinical and biochemical hyperandrogenism with normal ovulatory cycles and normal ovarian morphology.
2. Combined oral contraceptive pill indication for treatment: i) hyperandrogenism-related dermo-cosmetic complaints with psychoemotional impact; ii) endometrial protection; and/or iii) contraception desire.
3. Scheduled phlebotomy acceptation if randomly allocated.
4. Signed informed consent.

Exclusion Criteria:

1. Contraindication for blood donation.
2. Plasma ferritin < 76 pmol/l and/or transferrin saturation percent < 15%.
3. Anemia (plasma hemoglobin < 12 g/dl or hematocrit < 36%).
4. Chronic kidney disease (eGFR < 60 ml/min per 1.73 m2).
5. Personal history of dyslipidemia, hypertension, prediabetes, diabetes mellitus, gestational diabetes or cardiovascular events.
6. Treatment with oral contraceptives, antiandrogens, insulin sensitizers, drugs that might interfere with blood pressure regulation, lipid profile or carbohydrate metabolism, and oral/parenteral iron therapy for the previous 3 months to inclusion.
7. Previous surgical treatment for PCOS.
8. History of blood donation for the previous 12 months to inclusion.
9. Current history of infectious disease, inflammatory disease, liver disease, neurologic disease or malignancy.
10. Eating disorders. Body mass index < 18.5 Kg/m2.
11. Hereditary hemochromatosis.
12. Celiac disease or malabsorptive disorder.
13. Contraindication for treatment with combined oral contraceptives.
14. Pregnancy.
15. Current smoking, recreational drug use or excessive alcohol consumption (> 40 g per day).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Change in the Matsuda index from the circulating glucose and insulin concentrations during and standard oral glucose tolerance test. | one year
Percentage of patients with Hb < 12 g/dl or hematocrit <36% throughout the study | one year

SECONDARY OUTCOMES:
Change in the percentage of patients with undiagnosed prediabetes/diabetes between month 0 and 12 of follow-up | one year
Change in the Disposition index between month 0 and 12 of follow-up | one year
Change in the lipid profile between month 0 and 12 of follow-up | one year
Changes in the blood pressure recordings between month 0 and 12 of follow-up | one year
Percentage of patients with ferropenia throughout the study | one year
Percentage of patients with a hypovolemic event during blood donation | one year

OTHER OUTCOMES:
Subclinical chronic inflammation | one year
Oxidative stress | one year
Autonomic vascular function | one year
Blood clotting test | one year

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Luque Ramírez, M.D., Ph.D., Principal Investigator — Assistant in Endocrinology. Member of the Diabetes, Obesity and Human Reproduction Research Group from the lnstituto Ramón y Cajal de Investigación Sanitaria (IRYCIS)
Locations (1):
- Diabetes, Obesity and Human Reproduction Research Group, Department of Endocrinology and Nutrition, Hospital Universitario Ramón y Cajal, Universidad de Alcalá, Instituto Ramón y Cajal de Investigación Sanitaria (IRYCIS), Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
All data sets generated during and/or analyzed during the current study are not publicly available but are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: With publication
Access Criteria: Data are available from PI on reasonable request (manuel.luque@salud.madrid.org)

REFERENCES:
- [Result] Ortiz-Flores AE, Martinez-Garcia MA, Nattero-Chavez L, Alvarez-Blasco F, Fernandez-Duran E, Quintero-Tobar A, Escobar-Morreale HF, Luque-Ramirez M. Iron Overload in Functional Hyperandrogenism: In a Randomized Trial, Bloodletting Does Not Improve Metabolic Outcomes. J Clin Endocrinol Metab. 2021 Mar 25;106(4):e1559-e1573. doi: 10.1210/clinem/dgaa978. PMID 33462622
- [Result] Luque-Ramirez M, Ortiz-Flores AE, Nattero-Chavez L, Martinez-Garcia MA, Insenser M, Alvarez-Blasco F, Fernandez-Duran E, Quintero-Tobar A, de Lope Quinones S, Escobar-Morreale HF. Bloodletting has no effect on the blood pressure abnormalities of hyperandrogenic women taking oral contraceptives in a randomized clinical trial. Sci Rep. 2021 Nov 11;11(1):22097. doi: 10.1038/s41598-021-01606-7. PMID 34764381
- [Result] Luque-Ramirez M, Ortiz-Flores AE, Martinez-Garcia MA, Insenser M, Quintero-Tobar A, De Lope Quinones S, Fernandez-Duran E, Nattero-Chavez ML, Alvarez-Blasco F, Escobar-Morreale HF. Effect of Iron Depletion by Bloodletting vs. Observation on Oxidative Stress Biomarkers of Women with Functional Hyperandrogenism Taking a Combined Oral Contraceptive: A Randomized Clinical Trial. J Clin Med. 2022 Jul 3;11(13):3864. doi: 10.3390/jcm11133864. PMID 35807149